CLINICAL TRIAL: NCT04291781
Title: Phase II Clinical Trial of RC18(Recombinant Human B Lymphocyte Stimulator Receptor - Antibody Fusion Protein for Injection) in the Treatment of Primary IgA Nephropathy
Brief Title: A Study of RC18 Administered Subcutaneously to Subjects With Primary IgA(Immunoglobulin A) Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18C014
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — RC-18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RC18 160mg (Experimental): RC18 160mg subcutaneous injection (S.C.) once weekly ,and a total of 24 doses
  Interventions: Biological: RC18 160mg
- RC18 240mg (Experimental): RC18 240mg S.C. once weekly ,and a total of 24 doses
  Interventions: Biological: RC18 240mg
- Placebo (Placebo Comparator): Placebo S.C. once weekly ,and a total of 24 doses
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: RC18 160mg — subcutaneous injection on the upper arm, abdomen, or upper thigh outside;
  Other Names: Tai Ai, Recombinant Human B-Lymphocyte Stimulator Receptor- Antibody Fusion Protein
  Arms: RC18 160mg
Biological: RC18 240mg — subcutaneous injection on the upper arm, abdomen, or upper thigh outside;
  Other Names: Tai Ai, Recombinant Human B-Lymphocyte Stimulator Receptor- Antibody Fusion Protein
  Arms: RC18 240mg
Biological: placebo — subcutaneous injection on the upper arm, abdomen, or upper thigh outside;
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of Tai Ai(Recombinant Human B Lymphocyte Stimulator Receptor-Antibody Fusion Protein for Injection) in the treatment of IgA nephropathy.

DETAILED DESCRIPTION:
Both RC18 and Recombinant Human B Lymphocyte Stimulator Receptor-Antibody Fusion Protein for Injection are other names of Tai Ai.

After a 35-day screen period, subjects are randomly allocated into 3 groups receiving subcutaneous injection of Tai Ai 160mg, Tai Ai 240mg, and placebo once a week individually. The treatment lasts 24 weeks. Subjects, the sponsor, investigators are blinded in the whole process of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Signing the informed consent;
2. Biopsy confirmed diagnosis of IgA nephropathy;
3. Male or female, between 18 and 70 years age;
4. During screening, 24-hour urine protein excretion ≥0.75 g/24h at Visit 1 and/or Visit 2 and at Visit 3;
5. Estimated glomerular filtration rate (eGFR) (CKD-EPI ) >35 ml/min per 1.73m^2;
6. Have received the Angiotension converting enzyme Inhibitors(ACEI)/Angiotensin receptor blocker(ARB) standard treatment for 12 weeks prior to randomization, and have stabled the dosage (within the maximum tolerated dosage) for 4 weeks prior to randomization.

Exclusion Criteria:

1. Abnormal laboratory tests;
2. Any secondary IgA nephropathy caused by Henoch-Schönlein purpura, ankylosing spondylitis, systemic lupus erythematosus, sjogren syndrome, viral hepatitis, liver cirrhosis, rheumatoid arthritis, mixed connective tissue disease, polyarteritis nodosa, erythema nodosum, psoriasis, ulcerative colitis, crohn's disease, tumor, AIDS ,etc.;
3. Any nephropathy with special pathologic or clinical types, such as nephrotic syndrome, crescentic glomerulonephritis(with >50% of biopsied glomeruli), minimal change disease with IgA deposition; and IgA nephropathy requiring corticosteroids treatment.
4. Suffering from cardiovascular and cerebrovascular events (myocardial infarction, unstable angina, ventricular arrhythmia, New York heart association grade III-IV heart failure, stroke, etc.) within the last 12 weeks;
5. Treating with systemic corticosteroids drug(excluding topical or nasal steroids) within 3 months prior to randomizing;
6. Treating with systemic immunosuppressor within 3 months prior to randomizing: cyclophosphamide, azathioprine, mycophenolate mofetil, leflunomide, tacrolimus, cyclosporine, rituximab, tripterygium wilfordii, etc.;
7. Requiring hospitalization or intravenous antibiotics treatment due to active infection within 3 months prior to randomizing;
8. Active tuberculosis or latent carrier without treatment;
9. Herpes zoster infected patients or patients with positive HIV antibody or positive HCV antibody;
10. Active hepatitis or severe liver disease, and HBV infection (According to the HBV screening test, ① the HBsAg-positive; ②HBsAg-negative and HBcAb-positive, the HBV-DNA should be tested to determine the situation: the HBV-DNA positive subjects should be excluded, while the HBV-DNA negative subjects can participated in.)
11. With malignant tumors;
12. Pregnancy ，lactation, or patients with childbearing plans during the trial;
13. Nephrotoxic drugs is unavoidable during the study period;
14. Allergy to human-derived biologics;
15. Receiving any other investigating drug 4 weeks or 5 times half-life of the experimental drug (whichever is longer) prior to randomization;
16. Not suitable for the study judged by investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24-hour urine protein excretion at Week 24; | week 24
  based on the 24 -hour urine collection

SECONDARY OUTCOMES:
Change from baseline in estimated Glomerular Filtration Rate(eGFR) | week 0, 4, 8, 12, 16, 20, 24
  eGFR is calculated using the CKD-EPI method.
Change from baseline in urine protein/creatine ratio(UPCR) and/or urine albumin/ creatine ratio(UACR) | week 0, 4, 8, 12, 16, 20, 24
Change from baseline in Immunoglobulin G(IgG); | week 0, 4, 8, 12, 16, 20, 24
Change from baseline in Immunoglobulin M(IgM); | week 0, 4, 8, 12, 16, 20, 24
Change from baseline in Immunoglobulin A(IgA); | week 0, 4, 8, 12, 16, 20, 24
Change from baseline in the count of urine red blood cells | week 0, 4, 8, 12, 16, 20, 24
Change from baseline in the count of B-lymphocytes (CD19+) | week 0, 4, 8, 12, 16, 20, 24
Change from baseline in complement 3（C3） | week 0, 4, 8, 12, 16, 20, 24
Change from baseline in complement 4 (C4) | week 0, 4, 8, 12, 16, 20, 24
The incidence rate and severity of adverse events. | week 0, 4, 8, 12, 16, 20, 24
  An adverse event is any undesirable experience associated with the use of a medical product in a patient.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, M.D., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital., Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639